CLINICAL TRIAL: NCT04582786
Title: A Proof of Concept Randomized, Double-blind, Parallel Group, Controlled Dose-finding and Safety Study of STR-324 in Post-operative Pain
Brief Title: Dose Finding Study of STR-324
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alaxia SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STR-324-CL-072; 2019-003019-80 (EudraCT Number)
Record Dates: First submitted 2020-09-25; First posted 2020-10-12 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Step 1 of the study is single blinded for participants only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard group (Active Comparator): Standard treatment (morphine) administered according to usual practice
  Interventions: Drug: Morphine
- Test group: Infusion with bolus (Experimental): STR-324 or morphine HCl infusion started with a initial bolus
  Interventions: Drug: Morphine HCl; Drug: STR-324
- Test group: Infusion without bolus (Experimental): STR-324 or morphine HCl infusion started without a initial bolus
  Interventions: Drug: Morphine HCl; Drug: STR-324

INTERVENTIONS:
Drug: Morphine — Repeated bolus according to pain score
  Arms: Standard group
Drug: Morphine HCl — Infusion of morphine HCl solution for intravenous administration
  Arms: Test group: Infusion with bolus; Test group: Infusion without bolus
Drug: STR-324 — Infusion of solution for intravenous administration
  Arms: Test group: Infusion with bolus; Test group: Infusion without bolus

SUMMARY:
This study aims to evaluate the analgesic effect and the safety of 4 doses of STR-324 administered as an infusion, with or without initial bolus, to patients suffering from post-operative pain.

The sensitivity of the pain model used in the trial will be evaluated with a standard group treated with morphine under the usual care conditions.

DETAILED DESCRIPTION:
The first step (single-blind standard group) aims to verify the sensitivity of the study pain model in the proposed surgery to confirm the validity of the surgery according to their pain and enrolment rate. 12 patients are planned to be enrolled.

The second step (dose-finding study) is a randomized, double-blind, parallel groups, controlled clinical trial involving a total of 106 patients divided into two groups in which patients will be randomized between STR-324 and morphine HCl:

* Group 1: Titration initiated with a bolus
* Group 2: Titration without initial bolus.

ELIGIBILITY:
Selection criteria:

1. Patient aged ≥18 to <65 years old, at screening;
2. Having signed an informed consent prior to any study-related procedure;
3. Patients planned to undergo a major laparoscopic abdominal or pelvic surgery;
4. Surgery to be performed without local or regional anaesthesia nor infiltration;
5. Body mass index (BMI) between 18 and 30 kg/m² inclusive at screening, and with a minimum weight of 50 kg;
6. Women of childbearing potential must agree to use at least one effective contraceptive method upon enrolment and for 1 cycle following the last dose of the investigational product.

Inclusion Criteria:

The criteria for definitive enrolment must be checked in the Post-Anaesthesia Care Unit (PACU) at the inclusion visit:

1. NRS-measured pain intensity ranging from 4 to 8 inclusive at baseline PACU measurement;
2. With a sedation score ≤ S1 (awake or intermittently sleepy) at the time of pain assessment.

Exclusion Criteria:

1. Patient contra-indicated for morphine administration;
2. Unstable or poorly controlled psychiatric condition (e.g., untreated PTSD, major anxiety, or depression). Subjects who take stable doses (same dose >30 days) of antidepressants and/or anti-anxiety drugs may be included;
3. Women who are pregnant or breastfeeding;
4. History of alcohol, opiate or other drug abuse.
5. Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment might interfere with the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator. Minor deviations of values from the normal range may be accepted, if judged by the Investigator to have no clinical relevance;
6. Clinically significant abnormalities, as judged by the investigator, in laboratory test results;
7. Participation in an investigational drug or device study within 1 month prior to dosing.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative Change of Pain Intensity | On and/or after study drug, with fixed timepoints at 5, 10, 15, 20, 30, 45, 60, 75, 90, 105 and 120 minutes. If re-titration is required/performed, additional 5-minutes interval timepoints shall be added.
  Pain Intensity will be assessed by a Numerical Rating Scale (NRS) before and during analgesic infusion. Change of Pain Intensity assessed by the Numerical Rating Scale (NRS) after initiation of the post-op analgesia and before switch to standard treatment.
  The following parameter will be assessed:
  - Qualitative: a decrease of 2 units minimum from baseline and/or achievement of a pain score ≤ 3 is considered successful, responder=Yes.
Quantitative Change of Pain Intensity | On and/or after study drug, with fixed timepoints at 5, 10, 15, 20, 30, 45, 60, 75, 90, 105 and 120 minutes. If re-titration is required/performed, additional 5-minutes interval timepoints shall be added.
  Pain Intensity will be assessed by a Numerical Rating Scale (NRS) before and during analgesic infusion. Change of Pain Intensity assessed by the Numerical Rating Scale (NRS) after initiation of the post-op analgesia and before switch to standard treatment.
  The following parameter will be assessed:
  - Quantitative: maximum value of the pain score difference versus baseline.

SECONDARY OUTCOMES:
Adverse events collection | AEs collected directly after surgery until at least 30 days after the day of surgery.
  Any untoward medical occurrence in a patient or a clinical investigation subject, which does not necessarily have a causal relationship with the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes